CLINICAL TRIAL: NCT01346644
Title: Study of Tolerance of an Infant Formula Supplemented With Lactobacillus Fermentum CECT5716
Brief Title: Safety of Lactobacillus Fermentum in Newborn Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Puleva Biotech (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: P024
Record Dates: First submitted 2011-05-01; First posted 2011-05-03 (Estimated); Last update posted 2013-05-16 (Estimated); Status verified 2013-05

CONDITIONS: Tolerance
Keywords: Probiotic; infant nutrition; safety; infections
MeSH Terms: conditions — Infections | interventions — Infant Formula

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- No probiotics (Active Comparator): Infant formula with no probiotics
  Interventions: Other: Infant formula
- Probiotic (Experimental): Infant formula supplemented with probiotic
  Interventions: Other: Infant formula

INTERVENTIONS:
Other: Infant formula — Powder infant formula
  Arms: No probiotics
Other: Infant formula — Powder infant formula
  Arms: Probiotic

SUMMARY:
In the last years manipulation of intestinal microbiota with probiotics has gained an increasing interest, specially in infant nutrition since recent studies has demonstrated the presence of probiotics in human milk. However, there are few studies studying the effects of probiotics in newborns. The objective of the present study is to analyze safety and tolerance of the probiotic Lactobacillus fermentum CECT5716 isolated from human milk.

ELIGIBILITY:
Inclusion Criteria:

* Healthy 1 month infants exclusively formula-fed

Exclusion Criteria:

* gastrointestinal disorders (history of chronic diarrhoea or constipation, gastroesophageal reflux)
* gastrointestinal surgery
* cow's milk protein allergy
* metabolic disorders (diabetes, lactose intolerance)
* immune deficiency
* antibiotic prescription 1-week prior to inclusion and previous use of formula containing prebiotics or probiotics

Ages: 21 Days to 30 Days | Sex: All
Age Groups: Child
Enrollment: 137 (Actual)
Dates: Start 2009-02

PRIMARY OUTCOMES:
average weight gain | 4 months

SECONDARY OUTCOMES:
growth and health of infants | 2,4,6,12 and 36 months of life
  average weight, length of infants. Incidence of infections. Incidence of allergic diseases

CONTACTS AND LOCATIONS:
Overall Officials: Mercedes Gil, Doctor, Principal Investigator — Hospital Reina Sofía de Córdoba (Spain)
Locations (1):
- Biosearch Life, Granada, Granada, Spain

REFERENCES:
- [Derived] Maldonado-Lobon JA, Gil-Campos M, Maldonado J, Lopez-Huertas E, Flores-Rojas K, Valero AD, Rodriguez-Benitez MV, Banuelos O, Lara-Villoslada F, Fonolla J, Olivares M. Long-term safety of early consumption of Lactobacillus fermentum CECT5716: A 3-year follow-up of a randomized controlled trial. Pharmacol Res. 2015 May-Jun;95-96:12-9. doi: 10.1016/j.phrs.2015.01.006. Epub 2015 Feb 16. PMID 25697549